CLINICAL TRIAL: NCT01775709
Title: Evaluation of a New Biocompatible Pressure Equalizing Tube
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Hamid Djalilian, M.D.,Associate Professor of Clinical Otolaryngology, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20128774
Record Dates: First submitted 2013-01-14; First posted 2013-01-25 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Otitis Media
Keywords: middler ear infection
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PE tube with Duckbill Valve (Experimental): PE tube with Duckbill Valve
  Interventions: Device: PE tube with Duckbill Valve

INTERVENTIONS:
Device: PE tube with Duckbill Valve — PE tube with Duckbill Valve

SUMMARY:
Otitis media is the most common illness in children and 5% to 10% of their symptom cause by fluids in their middle ear . The OME can cause hearing loss included poor development of speech and poor communication.

The surgical procedure is considered simple and relatively safe, but several complications may occur after Pressure Equalizing tube insertion. The most prevalent complications are otorrhea, biofilm and formation of retraction pockets. Otorrhea occurs in 30% to 83% of children with tube and is mainly due bacterial contamination of the middle ear either from external ear canal or impaired Eustachian tube. Swimming can facilitate the entry of bacteria into the middle ear from the ear canal through the PE tubes, and this assumption is reinforced by the statistically significant association between the rate of otorrhea and the non-utilization of ear plugs in children who swim (from 47% in children who used ear plugs to 56% in those who did not).

DETAILED DESCRIPTION:
The researcher at Beckman Laser Institute, University of California, Irvine, develops new medical tool device call biocompatible Pressure Equalizing tube which can stop air passage and pressure equalization instantly, and can prevents water into the middle ear cavity. evaluate and compare the efficacy of a biocompatible Pressure Equalizing tube that enables air passage and pressure equalization almost instantly, while prevents the entrance of fluids, specially water, into the middle ear cavity.

The biocompatible Pressure Equalizing tube can reduce the rate of postoperative otorrhea,air passage between outside and middle ear cavity,prevents formation of retraction pockets in TM and swimming with lower risk of otorrhea.

ELIGIBILITY:
Inclusion Criteria:

1. Male/ female at all age- newborn to adult.
2. Non- pregnant woman.
3. Diagnose of middle ear infection and plan for surgery procedure

Exclusion Criteria:

1. Pregnant woman
2. Incompetent adults (i.e. individuals with cognitive impairment)
3. Presence of immunodeficiency; cystic fibrosis; sickle cell disease;
4. Another major systemic disease
5. Congenital malformation of the external, middle, or inner ear
6. Sensorineural hearing loss; otoneurologic disease
7. History of prior ear surgery such as tympanoplasty, tympanomastoidectomy, or mastoidectomy; cholesteatoma; chronic mastoiditis; intratemporal or intracranial suppurative complications of otitis media
8. Use of ototoxic medication (except topical use)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pressure-equalizing tube with Duckbill Valve stop air and water passage during middle ear infection treatment | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Botvinick, Ph.D., Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- UCIMC, Orange, California, United States